CLINICAL TRIAL: NCT01076192
Title: Post-authorization, Observational Study to Evaluate the Effectiveness of Adalimumab (HUMIRA®) on Moderate-severe Psoriasis Under Conditions of Routine Clinical Practice in Spain.
Brief Title: Study of Adalimumab (HUMIRA®) in Patients With Moderate to Severe Psoriasis (PS) in Spain (PROMISE)
Acronym: PROMISE
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: IMS Health (Other)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P11-067
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Moderate-to-severe Chronic Plaque Psoriasis
Keywords: Moderate Psoriasis; Psoriasis; Severe Psoriasis; Adalimumab; Effectiveness; Safety; Clinical practice
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Moderate-to-severe chronic plaque psoriasis: Participants with moderate-to-severe chronic plaque psoriasis treated with adalimumab in routine clinical practice

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of adalimumab as used in routine clinical practice in adult patients with moderate to severe chronic plaque psoriasis in Spain.

DETAILED DESCRIPTION:
PROMISE is a 2 year post-authorization study of patients taking adalimumab for Psoriasis. Patients who volunteer to participate will be asked to provide information about their medical history and experiences with adalimumab. No study specific testing will be performed. Patients will be asked to provide data on their experiences with adalimumab approximately every 6 months, or as determined by the study doctor. No drug will be provided as a result of participation in the registry. All treatment decisions are independent of participation in the registry. A total of 547 subjects were enrolled: 532 in the ITT population were analyzed for efficacy (excluding 15 for lack of follow-up visits (n=8), non-fulfillment of the criteria of moderate to severe PS (n=6) and failure to initiate treatment at the baseline visit (n=1)); 542 were analyzed for safety (excluding 5 due to lack of evaluable safety data).

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older.
* Patient diagnosed with moderate to severe chronic plaque PS beginning treatment with adalimumab in accordance with the authorized conditions of use.
* Patient gives informed consent in writing.

Exclusion Criteria:

* Patients who cannot be treated in accordance with the local product label
* Patient participating or going to participate in a clinical trial during the study follow-up
* Patient with difficulties for adequately reading, understanding and completing a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate-to-severe chronic plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2010-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Sancho Sanchez, PharmD, Study Director — Abbvie Farmaceutica, S.L.U. Spain

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 547 subjects were enrolled: 532 in the ITT population were analyzed for efficacy (excluding 15 for lack of follow-up visits (n=8), non-fulfillment of the criteria of moderate to severe PS (n=6) and failure to initiate treatment at the baseline visit (n=1)); 542 were analyzed for safety (excluding 5 due to lack of evaluable safety data).
Groups:
- Moderate-to-severe Chronic Plaque Psoriasis: Participants with moderate-to-severe chronic plaque psoriasis treated with Humira® in routine clinical practice
Period: Overall Study
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Started | 547
Completed | 350
Not Completed | 197
Not completed — Other | 197

BASELINE CHARACTERISTICS:
Population: Baseline analyses accounts for Intention to treat (ITT) population (all participants who received at least 1 dose of study drug and had at least 1 follow-up visit).
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 532
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.48 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 326

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI)
Description: PASI is a measurement of the severity of psoriasis. It is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A lower (and negative) value of change indicates an increase in the severity of the psoriasis, while a positive value indicates an improvement in the severity of the PS. Missing data were imputed using last observation carried forward (LOCF).
Time Frame: Baseline, month 1 and every 3 months the first year and every 6 months up to month 24
Population: Efficacy analyses included all participants who received at least 1 dose of adalimumab and had at least one follow-up visit (ITT) with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 528
units on a scale
  Month 1 | 8.39 (7.43)
  Month 3 | 11.30 (8.84)
  Month 6 | 11.52 (9.41)
  Month 9 | 11.32 (9.53)
  Month 12 | 11.21 (9.67)
  Month 18 | 10.93 (9.77)
  Month 24 | 10.91 (9.78)

2. Primary Outcome: Percentage of Participants Achieving a Reduction in PASI Score of at Least 50% (PASI 50)
Description: PASI is a measurement of the severity of psoriasis. It is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI 50 response is the percentage of participants who achieved at least a 50% reduction (improvement) from baseline in PASI score. Missing data were imputed using LOCF.
Time Frame: Baseline, month 1 and every 3 months the first year and every 6 months up to month 24
Population: Efficacy analyses included ITT population with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 526
percentage of participants
  Month 1 | 58.4
  Month 3 | 80.6
  Month 6 | 80.8
  Month 9 | 80.6
  Month 12 | 79.5
  Month 18 | 76.8
  Month 24 | 77.4

3. Primary Outcome: Percentage of Participants Achieving a Reduction in PASI Score of at Least 75% (PASI 75)
Description: PASI is a measurement of the severity of psoriasis. It is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI 75 response is the percentage of participants who achieved at least a 75% reduction (improvement) from baseline in PASI score. Missing data were imputed using LOCF.
Time Frame: Baseline, month 1 and every 3 months the first year and every 6 months up to month 24
Population: Efficacy analyses included ITT population with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 526
percentage of participants
  Month 1 | 29.8
  Month 3 | 64.8
  Month 6 | 66.9
  Month 9 | 65.8
  Month 12 | 64.6
  Month 18 | 63.7
  Month 24 | 64.4

4. Secondary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: DLQI is a self-administered Health Related Quality of Life (HRQL) questionnaire specifically for patients with dermatological diseases, adapted and validated in the Spanish population. It consists of 10 items with a Likert response scale for 4 categories and uses a 7 day time reference. It generates a global score that ranges from 0 (better HRQL) to 30 (worse HRQL) points. Change in DLQI was calculated by deducting the final score from the baseline score. Missing data were imputed using LOCF.
Time Frame: Baseline and every 6 months up to month 24
Population: Efficacy analyses included ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 504
units on a scale
  Month 6 | 5.83 (6.95)
  Month 12 | 6.17 (7.12)
  Month 18 | 6.05 (7.31)
  Month 24 | 5.99 (7.43)

5. Secondary Outcome: Mean Change From Baseline in EuroQol Quality of Life Questionnaire (EQ-5D) Visual Analogue Scale (VAS)
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where increased scores correspond to better HRQL. 0 is the 'worst imaginable health state' and 100 is the 'best imaginable health state'. Change in EQ-5D VAS score was calculated by deducting the final score from the baseline score. Increased scores correspond to better health state. Missing data were imputed using LOCF.
Time Frame: Baseline and every 6 months up to month 24
Population: Analysis included ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 453
units on a scale
  Month 6 | -10.79 (21.75)
  Month 12 | -12.27 (22.92)
  Month 18 | -12.91 (23.45)
  Month 24 | -12.71 (23.71)

6. Secondary Outcome: Mean Change From Baseline in Percentage of Lost Productivity Assessed Using Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI-SHP)
Description: WPAI-SHP is a questionnaire used to evaluate lost productivity. The scores on the WPAI questionnaire are presented as percentages (multiplying the scores by 100), with 0% representing no impact on productivity and 100% representing complete impact on productivity. Change in WPAI-SHP was calculated by deducting the final score from the baseline score. Increased (positive) scores correspond to a reduction in the percentage of lost work productivity. Missing data were imputed using LOCF. n=the number of participants with data at each time point.
Time Frame: Baseline and every 6 months up to month 24
Population: Analysis included ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale (a derived score)
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 251
units on a scale (a derived score)
  Month 6 (n=180) | 10.61 (24.97)
  Month 12 (n=145) | 9.86 (24.55)
  Month 18 (n=137) | 12.63 (25.39)
  Month 24 (n=121) | 12.89 (21.93)

7. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: AESIs are adverse events of special interest, including infection, neoplasm, lupus-like, demyelinating disease, serious hepatic and/or haematological event.
Time Frame: From time of informed consent to the final visit after 2 years of observation
Population: Analysis included safety analysis population i.e., all participants who received at least 1 dose of adalimumab with evaluable safety data.
Measure: Number; unit: participants
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 542
participants
  Cerebrovascular accident | 2
  Haematological event | 1
  Hepatic event | 1
  Congestive heart failure | 1
  Opportunistic infections | 30
  Lupus-like syndrome | 1
  Neoplasm | 11

8. Primary Outcome: Percentage of Participants Achieving a Reduction in PASI Score of at Least 90% (PASI 90)
Description: PASI is a measurement of the severity of psoriasis. It is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI 90 response is the percentage of participants who achieved at least a 90% reduction (improvement) from baseline in PASI score. Missing data were imputed using LOCF.
Time Frame: Baseline, month 1 and every 3 months the first year and every 6 months up to month 24
Population: Efficacy analyses included ITT population with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 526
percentage of participants
  Month 1 | 11.4
  Month 3 | 43.3
  Month 6 | 49.8
  Month 9 | 47.5
  Month 12 | 48.3
  Month 18 | 46.4
  Month 24 | 47.1

9. Primary Outcome: Percentage of Participants Achieving a Reduction in PASI Score of 100% (PASI 100)
Description: PASI is a measurement of the severity of psoriasis. It is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI 100 response is the percentage of participants who achieved a 100% reduction (improvement) from baseline in PASI score. Missing data were imputed using LOCF.
Time Frame: Baseline, month 1 and every 3 months the first year and every 6 months up to month 24
Population: Efficacy analyses included ITT population with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 526
percentage of participants
  Month 1 | 6.1
  Month 3 | 29.3
  Month 6 | 33.1
  Month 9 | 33.5
  Month 12 | 33.8
  Month 18 | 32.7
  Month 24 | 32.7

10. Primary Outcome: Mean Change From Baseline in Body Surface Area (BSA) Affected
Description: Body Surface Area (BSA) affected or the psoriasis area is determined by the direct calculation of the affected body surface area. This determination was used to evaluate the effectiveness of the treatment during each of the study visits. The change was calculated by deducting the final score from the baseline score. Increased scores correspond to reduction of severity and reduction of BSA. Missing data were imputed using LOCF.
Time Frame: Baseline, month 1 and every 3 months the first year and every 6 months up to month 24
Population: Efficacy analyses included ITT population with evaluable data.
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 509
percentage of body surface area
  Month 1 | 11.24 (15.51)
  Month 3 | 17.86 (18.43)
  Month 6 | 18.86 (19.58)
  Month 9 | 18.75 (19.73)
  Month 12 | 18.62 (19.63)
  Month 18 | 18.04 (19.76)
  Month 24 | 18.18 (20.08)

11. Primary Outcome: Percentage of Participants With Improvement From Baseline in Physician's Global Assessment (PGA)
Description: The PGA was used to measure participants' disease status at the time of assessment. This tool is a horizontal visual analogue 6-point scale measuring the degree of overall psoriatic lesion severity, and scores range from 0 (clear) to 5 (very severe). The percentage of patients who showed an improvement from baseline in their PGA scores is presented. Missing data were imputed using LOCF.
Time Frame: Baseline, month 1 and every 3 months the first year and every 6 months up to month 24
Population: Efficacy analyses included ITT population with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 530
percentage of participants
  Month 1 | 71.9
  Month 3 | 85.3
  Month 6 | 82.6
  Month 9 | 83.0
  Month 12 | 81.3
  Month 18 | 79.4
  Month 24 | 79.2

12. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs are adverse event with any of the following severity criteria: Potentially fatal/endangers life, Hospitalisation or prolonging of hospitalisation, a medically important event that requires medical or surgical intervention to prevent a serious outcome, Disability or persistent incapacitation, death, congenital anomalies and/or miscarriage or abortion.
  See the Reported Adverse Events Section for more details.
Time Frame: From time of informed consent to the final visit after 2 years of observation
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Number analyzed (Participants) | 542
participants | 24

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of study (Month 0) through month 24 following the start of treatment with adalimumab.
Description: Analysis included safety analysis population i.e., all participants who received at least 1 dose of adalimumab with evaluable safety data.
Arm/Group | Moderate-to-severe Chronic Plaque Psoriasis
Serious Adverse Events (participants affected / at risk) | 24/542
Other Adverse Events (participants affected / at risk) | 314/542
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate-to-severe Chronic Plaque Psoriasis (N=542)
Myelodisplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage of the digestive tract (Gastrointestinal disorders) | 2
Death (General disorders) | 1
Ferropenic anaemia (Blood and lymphatic system disorders) | 1
Lacunar stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Generalized weakness (General disorders) | 1
Hypertension (Vascular disorders) | 2
Vertigo (Nervous system disorders) | 1
Tuberculous meningitis (Infections and infestations) | 1
acute pancreatitis (Gastrointestinal disorders) | 1
outbreak of psoriasis (Skin and subcutaneous tissue disorders) | 2
subarachnoid haemorrhage after traumatic injury without mention of open intracraneal wound (Nervous system disorders) | 1
ureterohydronephrosis (Renal and urinary disorders) | 1
basocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
squamous cell carcinoma of the lungs (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
tonsil hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
scrotal abscess (Infections and infestations) | 1
clear cell carcinoma of the kidneys (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
chest pain (General disorders) | 1
arterial hypertension (Vascular disorders) | 2
myocardial infarction (Cardiac disorders) | 1
class iii heart failure (Cardiac disorders) | 1
neurosensory hypoacusia (Nervous system disorders) | 1
unstable angina (Cardiac disorders) | 1
psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 3
salmonellosis (Infections and infestations) | 1
astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
invasive breast duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
arthrodesis of the toe (Surgical and medical procedures) | 1
facial paralysis (Nervous system disorders) | 1
alcoholic pancreatitis (Gastrointestinal disorders) | 1
cardiac ablation (Surgical and medical procedures) | 1
non-specific tachycardia (Cardiac disorders) | 1
acute gastric ulcer with haemorrhage (Gastrointestinal disorders) | 1
angioedema (Skin and subcutaneous tissue disorders) | 1
spondylarthropathy (Musculoskeletal and connective tissue disorders) | 1
psoriatic arthopathy (Musculoskeletal and connective tissue disorders) | 2
ovarian benign germ cell teratoma (Reproductive system and breast disorders) | 1
suppurative hydradenitis (Skin and subcutaneous tissue disorders) | 1
sebaceous cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
complete auriculoventricular blockage (Cardiac disorders) | 1
allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1
multiorganic failure (General disorders) | 1
malignant neoplasms of the sigmoid colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
adenocarcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
state of confusion (Psychiatric disorders) | 1
tension headache (Nervous system disorders) | 1
non-specific chest pain (General disorders) | 1
deep vein thrombosis (Vascular disorders) | 1
hepatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
adenocarcinoma of the colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
radical prostatectomy (Surgical and medical procedures) | 1
abortion (Surgical and medical procedures) | 2
unwanted pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
community-acquired pneumonia (Infections and infestations) | 2
sarcoidosis (Immune system disorders) | 1
tonsillectomy (Surgical and medical procedures) | 1
peritonsillar abscess (Infections and infestations) | 1
worsening of psoriasis (Skin and subcutaneous tissue disorders) | 1
exacerbation of copd (Respiratory, thoracic and mediastinal disorders) | 1
septic arthritis (Musculoskeletal and connective tissue disorders) | 1
lupus-like syndrome (Immune system disorders) | 1
steroid-induced diabetes (Metabolism and nutrition disorders) | 1
pulmonary tuberculosis (Infections and infestations) | 1
sepsis caused by methicillin-resistant staphylococcus aureus (Infections and infestations) | 1
autoimmune hepatitis (Immune system disorders) | 1
infection by cytomegalovirus (Infections and infestations) | 1
miscarriage (Pregnancy, puerperium and perinatal conditions) | 1
ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
chrohn ileocolitis (Gastrointestinal disorders) | 1
adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
bronchial carcinoma, stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
leukocytosis (Blood and lymphatic system disorders) | 1
lymphocytosis (Blood and lymphatic system disorders) | 1
hysterectomy (Surgical and medical procedures) | 1
anxiety (Psychiatric disorders) | 1
vertigo syndromes and non-specific labyrinth disorders (Ear and labyrinth disorders) | 1
erysipela (Infections and infestations) | 1
chronic myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
carcinoma with unknown primary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
cervical lymphadenopathy (Blood and lymphatic system disorders) | 1
bacterial pyelonephritis (Infections and infestations) | 2
motorcycle accident (Injury, poisoning and procedural complications) | 1
comminuted fracture (Injury, poisoning and procedural complications) | 1
dislocated hip (Injury, poisoning and procedural complications) | 1
femur fracture (Musculoskeletal and connective tissue disorders) | 1
torn anterior cruciate ligament (Injury, poisoning and procedural complications) | 1
bariatric surgery (Surgical and medical procedures) | 1
septic shock (Infections and infestations) | 1
acute myocardial infarction of the inferoposterior wall (Cardiac disorders) | 1
pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
urothelial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
lung metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
bone metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
respiratory infection (Infections and infestations) | 1
infection by Escherichia coli (Infections and infestations) | 1
enterococcus bacteraemia (Infections and infestations) | 1
septicaemia by candida (Infections and infestations) | 1
normal nuclear magnetic resonance imaging (Investigations) | 1
oesophageal erosion (Gastrointestinal disorders) | 1
hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate-to-severe Chronic Plaque Psoriasis (N=542)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain not otherwise specified (Gastrointestinal disorders) | 2
Abnormal cholesterol in blood (Investigations) | 1
Abnormal gamma-glutamyl transferase (Investigations) | 2
Abnormal glucose (Investigations) | 1
Abnormal glutamate-pyruvate transaminase (Investigations) | 2
Abnormal uric acid in blood (Investigations) | 1
Abnormal erythrocytes (Blood and lymphatic system disorders) | 1
Abnormal menstruation (Reproductive system and breast disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Abnormal triglycerides (Investigations) | 1
Abnormal triglycerides in blood (Investigations) | 1
Abscess on a limb (Infections and infestations) | 1
Abscess on the back (Infections and infestations) | 1
Achilles tendinitis (Musculoskeletal and connective tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 4
Acute ear infection (Infections and infestations) | 2
Acute gastroenteritis (Gastrointestinal disorders) | 2
Acute pharyngitis (Infections and infestations) | 3
Acute sinusitis (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 9
Acute urticaria (Skin and subcutaneous tissue disorders) | 1
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Allergic reaction (Immune system disorders) | 1
Allergy to insect stings (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Anal pain (Gastrointestinal disorders) | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ankle pain (Musculoskeletal and connective tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 2
Anxiety attack (Psychiatric disorders) | 2
Arm pain (Musculoskeletal and connective tissue disorders) | 1
Arterial hypertension (Vascular disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 2
Articular inflammation (Musculoskeletal and connective tissue disorders) | 1
Asthenia (General disorders) | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Asthmatic bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Athlete's foot (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Average corpuscle volume (Investigations) | 1
Axillary abscess (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Balanitis (Reproductive system and breast disorders) | 1
Basocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Biliar colic (Hepatobiliary disorders) | 1
Blepharitis (Eye disorders) | 1
Boil (Infections and infestations) | 3
Bone fissure (Injury, poisoning and procedural complications) | 1
Bone oedema (Musculoskeletal and connective tissue disorders) | 1
Bronchiolitis caused by respiratory syncytial virus (Infections and infestations) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5
Cervical pain (Musculoskeletal and connective tissue disorders) | 1
Cervical lymphadenopathy (Blood and lymphatic system disorders) | 2
Cervicalgia (Musculoskeletal and connective tissue disorders) | 1
Chest pain (General disorders) | 1
Chest pain during exertion (Cardiac disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Chronic hepatitis C (Hepatobiliary disorders) | 1
Chronic nodular chondrodermatitis helicis (Ear and labyrinth disorders) | 1
Chronic renal insufficiency (Renal and urinary disorders) | 1
Circumcision (Surgical and medical procedures) | 1
Cold (Infections and infestations) | 20
Common cold (Infections and infestations) | 3
Common cold syndrome (Infections and infestations) | 2
Compressive neuropathy (Nervous system disorders) | 1
Condylomata (Infections and infestations) | 1
Condylomata acuminata (Infections and infestations) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Coronary artery calcification (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Cutaneous erythema (Skin and subcutaneous tissue disorders) | 1
Decline (Psychiatric disorders) | 1
Decompensated heart failure (Cardiac disorders) | 1
Decompensated diabetes (Metabolism and nutrition disorders) | 1
Decreased platelets (Investigations) | 2
Deficit of vitamin B12 (Metabolism and nutrition disorders) | 1
Dental fracture (Injury, poisoning and procedural complications) | 1
Dental implant (Surgical and medical procedures) | 1
Dental infection (Infections and infestations) | 5
Depression (Psychiatric disorders) | 1
Determination of C1Q (Investigations) | 1
Diabetes mellitus Type-2 (Metabolism and nutrition disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Dishydrotic eczema (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dorsalgia (Musculoskeletal and connective tissue disorders) | 1
Drowsiness (Nervous system disorders) | 1
Drug-induced liver disease (Hepatobiliary disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Dyspnea (Cardiac disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Earache (Ear and labyrinth disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Eczema of the eyelids (Skin and subcutaneous tissue disorders) | 1
Elevated alpha-fetoprotein (Investigations) | 1
Elevated amylase (Investigations) | 1
Elevated average corpuscle volume (Investigations) | 1
Elevated creatinine (Investigations) | 1
Elevated ferritin in plasma (Investigations) | 1
Elevated glutamate oxaloacetate transaminase (Investigations) | 1
Elevated glutamate-pyruvate transaminase (Investigations) | 5
Elevated high-density lipoprotein (Investigations) | 1
Elevated lipase (Investigations) | 1
Elevated triglycerides (Investigations) | 6
Elevated gammaglobulin (Investigations) | 1
Elevated transaminases (Investigations) | 5
Elevation of creatine phosphokinase (Investigations) | 1
Elevation of gamma-glutamyl transferase (Investigations) | 1
Enthesitis (Musculoskeletal and connective tissue disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 2
Epidermal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Epididimoorquitis (Reproductive system and breast disorders) | 1
Epigastralgia (Gastrointestinal disorders) | 3
Epigastric pain (Gastrointestinal disorders) | 1
Epileptic crisis (Nervous system disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erectile impotence (Reproductive system and breast disorders) | 1
Erosive gastritis (Gastrointestinal disorders) | 1
Exacerbation of psoriasis (Skin and subcutaneous tissue disorders) | 1
Excessive tearing (Eye disorders) | 1
Exhaustion (General disorders) | 1
Extraction of wisdom tooth (Surgical and medical procedures) | 1
Eye discomfort (Eye disorders) | 1
Face cellulitis (Infections and infestations) | 1
Facial paralysis (Nervous system disorders) | 1
Facial rash (Skin and subcutaneous tissue disorders) | 1
Falls (Injury, poisoning and procedural complications) | 5
Ferropenic anaemia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Flu (Infections and infestations) | 13
Foot cellulitis (Infections and infestations) | 2
Foot pain (Musculoskeletal and connective tissue disorders) | 1
Fractured metatarsal (Injury, poisoning and procedural complications) | 1
Functional dyspepsia (Gastrointestinal disorders) | 1
Furunculosis (Infections and infestations) | 2
Gastritis caused by helicobacter pylori (Infections and infestations) | 1
Gastroenteritis (Gastrointestinal disorders) | 2
General discomfort (General disorders) | 3
Generalised rash (Skin and subcutaneous tissue disorders) | 1
Genital candidiasis (Infections and infestations) | 2
Genital wart (Infections and infestations) | 2
Gingivitis (Gastrointestinal disorders) | 1
Glare (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Gonalgia (Musculoskeletal and connective tissue disorders) | 1
Granulomatous lesion (Skin and subcutaneous tissue disorders) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 7
Heel pain (Musculoskeletal and connective tissue disorders) | 1
Heel spur (Musculoskeletal and connective tissue disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 5
Herniated disc (Musculoskeletal and connective tissue disorders) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
High cholesterol (Investigations) | 9
Hormonal imbalance (Investigations) | 1
Hydrocele (Reproductive system and breast disorders) | 1
Hypercholesterolemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypertension attack (Vascular disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12
Hyperuricemia (Metabolism and nutrition disorders) | 4
Hypothyroidism (Endocrine disorders) | 1
Increase in size of submaxillar gland (Gastrointestinal disorders) | 1
Increased low-density lipoprotein (Investigations) | 2
Increased C-Reactive Protein (Investigations) | 1
Increased average corpuscular haemoglobin (Investigations) | 1
Increased bilirubin (Investigations) | 2
Increased creatine phosphokinase (Investigations) | 1
Increased gamma-glutamyl transferase (Investigations) | 4
Increased rheumatoid factor (Investigations) | 1
Increased serum glutamate-pyruvate transaminase (Investigations) | 3
Increased urea in blood (Investigations) | 1
Increased Hepatitis B viral load (Investigations) | 1
Increased vertical sleeve gastrectomy (Investigations) | 3
Ineffective drug (General disorders) | 1
Infected cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Infected sebaceous cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infection by blastocystis hominis (Infections and infestations) | 1
Infection of upper airways not otherwise specified (Infections and infestations) | 17
Inflammation of the middle ear (Ear and labyrinth disorders) | 1
Inguinal abscess (Infections and infestations) | 1
Insomnia (Nervous system disorders) | 1
Instability (Nervous system disorders) | 1
Intestinal polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intoxication by immunosuppressants (Injury, poisoning and procedural complications) | 1
Irritable bowel (Gastrointestinal disorders) | 1
Irritation of the palate (Gastrointestinal disorders) | 1
Itching in the injection zone (General disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Joint paint with involvement of the lower leg (Musculoskeletal and connective tissue disorders) | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 1
Labial herpes (Infections and infestations) | 1
Latent tuberculosis (Infections and infestations) | 2
Leg cellulitis (Infections and infestations) | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Leukoplakia of the oral mucosa (incl. tongue) (Gastrointestinal disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Loss of dental piece (Gastrointestinal disorders) | 1
Low folic acid (Investigations) | 1
Lower back pain (Musculoskeletal and connective tissue disorders) | 5
Low-grade fever (General disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Lupus-like syndrome (Immune system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Macrocytosis (Blood and lymphatic system disorders) | 1
Maculopapular rash (Skin and subcutaneous tissue disorders) | 1
Mandibular osteomyelitis (Infections and infestations) | 1
Megaloblastic anaemia (Blood and lymphatic system disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Navicular fractures (Musculoskeletal and connective tissue disorders) | 1
Negative tuberculosis test (Investigations) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Non-specific chest pain (Infections and infestations) | 1
Non-specific middle ear function (Infections and infestations) | 1
Viral infection not otherwise specified (Infections and infestations) | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 2
Oedema of the face (General disorders) | 1
Oedema of the feet (General disorders) | 1
Oedema of the leg (General disorders) | 1
Oedema of the limbs (General disorders) | 1
Oedema of the lower limbs (General disorders) | 1
Onphalitis (Infections and infestations) | 1
Ophthalmological herpes simplex (Infections and infestations) | 1
Oral infection (Infections and infestations) | 1
Osteoarthrosis (Musculoskeletal and connective tissue disorders) | 1
Osteoarticular pain (Musculoskeletal and connective tissue disorders) | 2
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Outbreak of psoriasis (Skin and subcutaneous tissue disorders) | 27
Outer ear infection (Infections and infestations) | 1
Pain at the puncture location (General disorders) | 2
Pain in hand (Musculoskeletal and connective tissue disorders) | 2
Pain in lower limbs (Musculoskeletal and connective tissue disorders) | 1
Pain in molars (Gastrointestinal disorders) | 1
Pain in the injection zone (General disorders) | 1
Painful knees (Musculoskeletal and connective tissue disorders) | 1
Painful tongue (Gastrointestinal disorders) | 1
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 2
Palpitations (Cardiac disorders) | 1
Paradoxical reaction to a drug (General disorders) | 2
Paraesthesia in limbs (Nervous system disorders) | 4
Paronychia (Infections and infestations) | 1
Paroxistic tachycardia (Cardiac disorders) | 1
Penile candidiasis (Infections and infestations) | 1
Perianal abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 14
Pharyngitis not otherwise specified (Infections and infestations) | 1
Pharyngoamygdalitis (Infections and infestations) | 7
Phlebitis (Vascular disorders) | 1
Photocoagulation (Surgical and medical procedures) | 1
Photophobia (Eye disorders) | 1
Pneumonia (Infections and infestations) | 3
Polymenorrhea (Reproductive system and breast disorders) | 1
Polyuria (Renal and urinary disorders) | 3
Positive antinuclear antibodies (Investigations) | 9
Positive cutaneous tuberculosis test (Investigations) | 1
Positive lupus anticoagulant (Investigations) | 1
Positive tuberculosis test (Investigations) | 5
Posterior detachment of the vitreous humour (Eye disorders) | 1
Post-surgical pain (General disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Pseudopterigion (Eye disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Psoriasis guttata (Skin and subcutaneous tissue disorders) | 1
Psoriasis of the scalp (Skin and subcutaneous tissue disorders) | 1
Psoriatic arthopathy (Musculoskeletal and connective tissue disorders) | 3
Psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 7
Pulmonary consolidation (Respiratory, thoracic and mediastinal disorders) | 1
Purulent secretion (Infections and infestations) | 1
Raynaud's disease (Vascular disorders) | 1
Reaction at injection site (General disorders) | 3
Rectorrhage (Gastrointestinal disorders) | 1
Reduced sex drive (Psychiatric disorders) | 2
Renal colic (Renal and urinary disorders) | 5
Renal lithotripsy (Surgical and medical procedures) | 1
Respiratory infection (Infections and infestations) | 1
Rheumatic polymyalgia (Immune system disorders) | 1
Rib fracture (Musculoskeletal and connective tissue disorders) | 1
Root canal (Surgical and medical procedures) | 1
Sciatic (Nervous system disorders) | 2
Scrotal abscess (Infections and infestations) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Senile purpura (Vascular disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2
Sinusitis (Infections and infestations) | 4
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Sore left arm (Musculoskeletal and connective tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Sprained ankle (Musculoskeletal and connective tissue disorders) | 1
Stasis dermatitis (Vascular disorders) | 1
Stiffness in the morning (Musculoskeletal and connective tissue disorders) | 1
Stiffness of limbs (Musculoskeletal and connective tissue disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Streptococcus tonsillitis (Infections and infestations) | 1
Sudden deafness (Ear and labyrinth disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tarry stool (Gastrointestinal disorders) | 1
Telogen alopecia (Skin and subcutaneous tissue disorders) | 1
Tendinitis (Musculoskeletal and connective tissue disorders) | 1
Terrien's marginal degeneration (Eye disorders) | 1
Throbbing headache (Nervous system disorders) | 1
Thyroid node (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Tingling sensation (Nervous system disorders) | 1
Tooth abscess (Infections and infestations) | 2
Tooth extraction (Surgical and medical procedures) | 3
Tooth sensitivity (Gastrointestinal disorders) | 1
Traffic accident (Injury, poisoning and procedural complications) | 2
Transaminitis (Investigations) | 8
Trauma injuries of limbs (Injury, poisoning and procedural complications) | 1
Tubular colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Twisted and sprained feet (Musculoskeletal and connective tissue disorders) | 1
Unspecified intestinal parasitosis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 9
Urinary tract infection by Escherichia (Infections and infestations) | 1
Urination disorder (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Vaginal candidiasis (Infections and infestations) | 2
Verruca vulgaris (Infections and infestations) | 2
Vertigo (Ear and labyrinth disorders) | 1
Viral gastroenteritis (Infections and infestations) | 1
Viral rash (Infections and infestations) | 1
Viriasis (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 3
Vulvovaginal candidiasis (Infections and infestations) | 4
Warts (viral) (Infections and infestations) | 3
Weight gain (Investigations) | 3
Weight loss (Investigations) | 2
Worsening of crohn's disease (Gastrointestinal disorders) | 1
Worsening of the disease (General disorders) | 1
Worsening of depression (Psychiatric disorders) | 1
Worsening of psoriasis (Skin and subcutaneous tissue disorders) | 3
Wound infection (Infections and infestations) | 1
Xerophthalmia (Eye disorders) | 1
Hypersensitivity at injection site (General disorders) | 1
Traumatic injuries of the lumbosacral plexus (Injury, poisoning and procedural complications) | 1
Bradycardia (Cardiac disorders) | 1
Broken meniscus (Musculoskeletal and connective tissue disorders) | 1
Hypertensive nephropathy (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.